CLINICAL TRIAL: NCT04794608
Title: Hypnosis in Virtual Reality in Patients in Protector Isolation Room for Aplasia in Clinical Hematology. Monocentric, Comparative, Randomized, Open Study.
Brief Title: Hypnosis in Virtual Reality in Patients in Protector Isolation Room for Aplasia in Clinical Hematology.
Acronym: Hyp_Hem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Privé Sévigné (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A02561-38
Record Dates: First submitted 2021-03-03; First posted 2021-03-12 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Aplasia
Keywords: Aplasia; Anxiety; Hypnosis; Virtual reality; Protector isolation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HypnoVR Arm (Experimental): During the three days of study in protector isolation, patients benefit from a 20-minute session of medical hypnosis in virtual reality.
  Interventions: Device: HYPNO VR® device
- Control Arm (No Intervention): During the three days of study in protector isolation, patients benefit from a 20-minute session of activity among those currently proposed in the service of hematology (reading, music, television).

INTERVENTIONS:
Device: HYPNO VR® device — The HYPNO VR® device is a software application of medical hypnosis in the treatment of pain and anxiety. It is associated with equipment: a virtual reality headset and a headphone.
  Before each session of hypnosis, the nursing staff offers patients the choices: visual universe, musical theme, male or female voice. The nursing staff selects the program, selects a duration of 20 minutes and presses start to start the medical hypnosis session in virtual reality.
  After completing the hypnotic trance sequence, as in a classic session, the patient is brought back to the "return" and exit hypnosis phase under the supervision of the nursing staff.
  Arms: HypnoVR Arm

SUMMARY:
Hematology patients are frequently treated in hospital for aplasia. Patients are then placed in protective isolation room. This situation of protective isolation can represent a significant source of stress and anxiety for the patient. Hypnosis is already used to treat anxiety in patients with cancer.

The purpose of this study is to evaluate the impact of virtual reality medical hypnosis sessions on anxiety and chronic pain of patients hospitalized for aplasia in order to broaden the supportive care proposals in the clinical hematology service of Sévigné Private Hospital.

DETAILED DESCRIPTION:
After verifying the patient's eligibility criteria and obtaining the signed informed consent form, the patient is randomized to the arm receiving hypnosis in virtual reality or to the control arm. The study ends after three consecutive days in protector isolation with one session hypnosis in virtual reality per day.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years.
* Haematological pathology
* Patient hospitalized in protective isolation for aplasia defined by a rate of polymorphonuclear neutrophils <0.5 G / L.
* Patient having signed his informed consent.
* Patient with social security coverage.
* Patient treated and monitored in the center for the duration of the study (maximum 1 month)

Exclusion Criteria:

* Patient unable to undergo protocol monitoring for psychological, social, family or geographic reasons.
* Patient deprived of his liberty or under guardianship.
* Patient with an underlying or concomitant pathology incompatible with inclusion in the trial, whether psychiatric or somatic
* Patient with a contraindication to the use of virtual reality (psychiatric disorders, unbalanced epilepsy, visual or hearing disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Compare the change in anxiety in the HYPNOVR group versus the change in anxiety in the "selected activity" control group. | For up to 3 days, every days (before and after the virtual reality hypnosis sessions), starting on day of inclusion.
  Comparison of the change in the anxiety "state" by the State Trait Anxiety Inventory (STAI) - State score before (15 minutes) and after (15 minutes) each virtual reality hypnosis session for 3 consecutive days (ie six questionnaires) to the change in the anxiety "state" in patients in the control group (STAI-State score evaluated 15 minutes before and 15 minutes after the patient was offered an activity of his choice). The score is a quantitative variable with values ranging from 20 to 80. The higher the score is, the more important the anxiety is.

SECONDARY OUTCOMES:
Test the hypothesis that medical hypnosis in virtual reality is accompagnied by a variation of the chronic pain (in comparision with a control group). | For up to 3 days, every days (before and after the virtual reality hypnosis sessions), starting on day of inclusion.
  Comparison of the change in chronic pain before and after each hypnosis session for the Hypno VR group, for 3 consecutive days, i.e. six assessments, in comparison with change in chronic pain in patients in the control group (also six assessments). The scale used is the visual analogical scale of pain which comes in the form of a ruler on which a cursor can be moved from end to end (from "no pain" to "maximum imaginable pain"). The rear face of the ruler, intended for the evaluator, has a graduation from 0 to 100 mm. The higher the score is, the more important the pain is.
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a modification in the consumption of analgesic treatments (in comparision with a control group). | For up to 3 days, every days (record before the virtual reality hypnosis sessions), starting on day of inclusion.
  Comparison of the proportion of analgesic treatments consumption (posology stopped, added or changed) for each day of the study between the two arms.
Test the hypothesis that medical hypnosis in virtual reality is accompanied by a modification in the consumption of anxiolytics treatments (in comparision with a control group). | For up to 3 days, every days (record before the virtual reality hypnosis sessions), starting on day of inclusion.
  Comparison of the proportion of anxiolytics treatments consumption (posology stopped, added or changed) for each day of the study between the two arms.
Test the hypothesis that medical hypnosis in virtual reality is accompagnied by a good patient satisfaction regarding the use of the virtual reality headset. | For up to 3 days, every days (record after the virtual reality hypnosis sessions), starting on day of inclusion.
  Assessment of the overall satisfaction of the patient in the HYPNO VR group by the satisfaction questionnaire (ie a questionnaire after each hypnosis session for 3 consecutive days). A level of satisfaction (on a 11-point scale from 0 to 10) of the patient will be measure for the state of relaxation, security, understanding, overall satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Violaine DONCKER, MD, Principal Investigator — Hôpital Privé Sévigné
Locations (1):
- Hôpital Privé Sévigné, Cesson-Sévigné, France

IPD SHARING:
Plan to Share IPD: No